CLINICAL TRIAL: NCT04484064
Title: Optimization of Targeted Anticancer Therapies: a Systematic Collection and Modeling of Pharmacokinetic Data and Elaboration of an Adherence Program
Brief Title: Optimization of the Targeted Anticancer Therapies
Acronym: OpTAT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Collaborators: Center for Primary Care and Public Health (Unisante), University of Lausanne, Switzerland (Other); Krebsforschung Schweiz, Bern, Switzerland (Other)
Responsible Party: Principal Investigator, Chantal Csajka, Director and Professor of the Center for Research and Innovation in Clinical Pharmaceutical Sciences, Centre Hospitalier Universitaire Vaudois
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CHUV-PCL-OpTAT-2015; 65/15 (Other: CER-VD)
Record Dates: First submitted 2016-01-28; First posted 2020-07-23 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: Cancer
Keywords: Cancer; Medication adherence; Oral targeted anticancer drugs; Population pharmacokinetics; Pharmacodynamic-pharmacokinetics relationships
MeSH Terms: conditions — Neoplasms; Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard care (No Intervention): Patients in the "standard care" arm will use an electronic adherence monitor (MEMS®) without any feedback (electronic data will be blinded to patients, clinicians and investigators until the analysis)
- Adherence program (Experimental): Patients in the "adherence program" will use the MEMS® and the pharmacist will provide an electronic feedback on medication adherence since the last visit. The identified determinants of medication adherence will be discussed with the patient.
  Interventions: Behavioral: Adherence program

INTERVENTIONS:
Behavioral: Adherence program — This program combines adherence evaluation using an electronic monitor (MEMS®) and feedback with repeated medication adherence interviews with the pharmacist.
  Arms: Adherence program

SUMMARY:
The study includes an observational pharmacokinetic study and an interventional medication adherence study. The purpose of this study is 1) to describe the concentration-time profiles of targeted anticancer drugs and to characterize the concentration-effect/toxicity relationships in the target population of patients (observational study) and 2) to characterize patterns of adherence to oral targeted anticancer drugs and identify key-driver modifiable adherence factors in patients participating in an adherence program (interventional study).

DETAILED DESCRIPTION:
Targeted anticancer therapies are often prescribed at the same dosage regimen in all patients. However, it is known that the marked interindividual variability in drug level may affect treatment outcomes. Several factors are known to modulate drug levels, such as weight, genetics host-drug and drug-drug interaction. The identification of these factors could give the possibility to propose better adjusted dosage regimens according to patient's individual characteristics. Moreover, the presence of high or low drug concentrations may partially explain toxicity or lack of efficacy of targeted anticancer drugs in some patients. The characterization of the relationship between drug levels and treatment response (efficacy and toxicity) would allow an optimized and a more individualized patient management with targeted anticancer drugs.

Oral targeted therapies must be taken on the long term and adherence issues have been shown to compromise treatment efficacy. Side effects and lifestyle management are among factors affecting treatment adherence. The characterization of adherence over time and the identification of factors susceptible to improve it will represent a great benefit for healthcare professionals and patients.

ELIGIBILITY:
Inclusion Criteria:

* Cancer patients to whom a targeted anticancer therapy is prescribed

Exclusion Criteria:

* Patients incapable of judgment or participants under tutelage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2015-05; Primary Completion 2020-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Blood concentrations of targeted anticancer drugs | A maximum of 8 blood samples are collected within 2 years after the inclusion (at maximum 1 blood sample per month).
  During their medical visits, from 1 to 8 blood samples will be collected per patients at the same moment as routine blood sampling. Drug concentration will be measured by HPLC-MS/MS.
Apparition of adverse events of targeted anticancer drugs | Adverse events are monitored at each medical visit (once per month) from the inclusion in the study during 2 years maximum or from the inclusion in the study to the end of the treatment.
  Adverse events are assessed during the routine medical visits according the National Cancer Institute Common Toxicity Criteria (NCI-CTCAE scale).
Change from treatment start in efficacy of targeted anticancer drugs | The cancer progression is evaluated at each PET-scan (once per 3 months) from the inclusion in the study during 2 years maximum or from the inclusion in the study to the end of the treatment.
  The progression free survival (PFS) is used to evaluate the drug efficacy. The PFS is defined as the time interval between the first dose of drug and the date of progression or any cause death. Patient without progression at the study end will be censored.

SECONDARY OUTCOMES:
Medication adherence : persistence rate and daily implementation of targeted anticancer drugs | 12 months
  Adherence to oral anticancer therapies will be monitored thanks to Electronic monitoring Systems (MEMS, AARDEX) during maximum 12 months. This is a 1:1 randomized medication adherence intervention, which compares an intervention group vs. usual care. The intervention consists in monthly motivational interviewing sessions between the patient and the pharmacist, along with the delivering of oral targeted anticancer drugs in electronic pill bottles (Electronic Event Monitoring EEM, MEMSTM, AARDEX Ltd.). The patient meet the pharmacist after each clinical visits (usually once per month).

CONTACTS AND LOCATIONS:
Overall Officials: Chantal Csajka, PharmD, PhD, Principal Investigator — Clinical Pharmacy Sciences
Locations (1):
- CHUV, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bandiera C, Cardoso E, Locatelli I, Zaman K, Diciolla A, Digklia A, Stravodimou A, Cristina V, Aedo-Lopez V, Dolcan A, Sarivalasis A, Bouchaab H, Pasquier J, Dotta-Celio J, Peters S, Wagner D, Csajka C, Schneider MP. A pharmacist-led interprofessional medication adherence program improved adherence to oral anticancer therapies: The OpTAT randomized controlled trial. PLoS One. 2024 Jun 7;19(6):e0304573. doi: 10.1371/journal.pone.0304573. eCollection 2024. PMID 38848380
- [Derived] Bandiera C, Cardoso E, Locatelli I, Digklia A, Zaman K, Diciolla A, Cristina V, Stravodimou A, Veronica AL, Dolcan A, Sarivalasis A, Liapi A, Bouchaab H, Orcurto A, Dotta-Celio J, Peters S, Decosterd L, Widmer N, Wagner D, Csajka C, Schneider MP. Optimizing Oral Targeted Anticancer Therapies Study for Patients With Solid Cancer: Protocol for a Randomized Controlled Medication Adherence Program Along With Systematic Collection and Modeling of Pharmacokinetic and Pharmacodynamic Data. JMIR Res Protoc. 2021 Jun 29;10(6):e30090. doi: 10.2196/30090. PMID 34185020